CLINICAL TRIAL: NCT05387395
Title: Impact of COVID 19 Vaccination or Infection on Disease Activity in Radiologically Isolated Syndrome Cohort: the VaxiRIS Study
Brief Title: COVID-19 on Disease Activity in Radiologically Isolated Syndrome Cohort
Acronym: VaxiRIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Neuro02
Record Dates: First submitted 2022-05-23; First posted 2022-05-24 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis; COVID-19
MeSH Terms: conditions — Multiple Sclerosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- complete vaccination: Complete vaccination was defined as administering two doses of mRNA or AstraZeneca vaccine, administration of one dose of Jansen vaccine, or administration of one dose of any vaccine in patients with a history of COVID19 infection.
  Interventions: Other: NO intervention
- incomplete vaccination: Other cases were defined as incomplete or absent vaccination.
  Interventions: Other: NO intervention

INTERVENTIONS:
Other: NO intervention — no intervention

SUMMARY:
The Radiologically Isolated Syndrome (RIS) is defined as incidental Magnetic Resonance Imaging (MRI) abnormalities fulfil the criteria for dissemination in space, suggestive of multiple sclerosis. Nowadays, mandatory vaccination in patients with multiple sclerosis (MS) is widely recommended. Regarding COVID19, the absence of specific warnings led to the proposal of vaccination in patients with inflammatory diseases of the central nervous system. We aimed to evaluate if COVID19 vaccination or infection increased the risk of clinical conversion to multiple sclerosis or evidence of disease activity (EDA) in a cohort of RIS subjects.

ELIGIBILITY:
Inclusion Criteria:

* patients belong to the RISC cohort;
* totally vaccinated ou partially vaccinated patient
* vaccination status known

Exclusion Criteria:

* presented a first clinical event before the COVID19 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients fulfilling the Radiologic Isolated Syndrome criteria
Sampling Method: Non-Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
COVID 19 vaccination and clinical conversion to multiple sclerosis risk | year 2
  number of patients with a conversion to MS in each group

SECONDARY OUTCOMES:
COVID 19 vaccination and evidence disease activity risk | year 2
  number of patients with an evidence disease activity in each group
multiple sclerosis evolution and history of COVID 19 infection | year 2
  number of patients with a conversion to MS in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided